CLINICAL TRIAL: NCT02287688
Title: Post-licensure Observational Safety Surveillance Study of Quadrivalent Meningococcal ACWY Conjugate Vaccine MenACWY-CRM (MENVEO®) in Children 2 Months Through 23 Months of Age.
Brief Title: Meningococcal Quadrivalent CRM-197 Conjugate Vaccine Infant Study
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 205534; V59_74OB (Other: Novartis)
Record Dates: First submitted 2014-10-27; First posted 2014-11-11 (Estimated); Results first posted 2019-10-21 (Actual); Last update posted 2019-10-21 (Actual); Status verified 2019-10

CONDITIONS: Meningococcal Disease; Infections, Meningococcal
Keywords: safety of Meningococcal quadrivalent CRM-197 conjugate vaccine; Children 2-23 months of age
MeSH Terms: conditions — Meningococcal Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Exposure group: Subjects aged 2-23 months who received at least one dose of the MenACWY-CRM vaccine at a Kaiser Permanente Southern California (KPSC) facility while enrolled as a KPSC health plan member.
  Interventions: Biological: Meningococcal quadrivalent CRM-197 conjugate vaccine

INTERVENTIONS:
Biological: Meningococcal quadrivalent CRM-197 conjugate vaccine — This study is strictly observational. Decisions of vaccination are made by health care providers.

SUMMARY:
This safety surveillance study of GlaxoSmithKline's quadrivalent meningococcal ACWY conjugate vaccine (Meningococcal quadrivalent CRM-197) among children 2 months through 23 months of age is a post-marketing study required by the United States Food and Drug Administration.

It is an observational study of children 2-23 months of age who receive at least one dose of MenACWY-CRM vaccine at a Kaiser Permanente Southern California facility (KPSC) while enrolled as a KPSC health plan member.

The objective of the infant study is to describe medical events that require emergency room visit or hospitalization in 6 months following MenACWY-CRM vaccination in children 2-23 months of age in a health maintenance organization in the United States. Outcomes include medical events that require emergency room visits or hospitalizations in children 2-23 months of age following any dose of MenACWY-CRM vaccination. Events with a history of the same diagnosis prior to the first dose of MenACWY-CRM vaccination will be excluded as a pre-existing condition.

ELIGIBILITY:
Inclusion Criteria:

* children 2-23 months of age at the time of MenACWY-CRM vaccination
* hold KPSC membership at the time of MenACWY-CRM vaccination
* vaccinated with MenACWY-CRM during the study period in KPSC

Exclusion Criteria:

* None

Ages: 2 Months to 23 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children 2-23 months of age who receive at least one dose of MenACWY-CRM vaccine at a Kaiser Permanente Southern California (KPSC) facility while enrolled as a KPSC health plan member.
Sampling Method: Non-Probability Sample
Enrollment: 144 (Actual)
Dates: Start 2014-12-01 (Actual); Primary Completion 2017-11-29 (Actual); Study Completion 2017-11-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Pasadena, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: There were 5,612,052 members of Kaiser Permanente of Southern California (KPSC) health plan during the study period. Among these,108,325 were children 2 to 23 months old. A total of 144 subjects aged 2 to 23 months who received at least one dose of MenACWY-CRM vaccine, were enrolled in this study.
Pre-assignment Details: Out of the 144 subjects enrolled, only 138 subjects were analysed in this study as 6 subjects did not meet the inclusion criteria.
Period: Overall Study
Arm/Group | Exposure Group
Started | 138
Completed | 138
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Exposure Group
Number analyzed (Participants) | 138
Age, Continuous [Mean (Standard Deviation); unit: Months]
  Age at first vaccination | 11.5 (6.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Gender: Female | 70
  Gender: Male | 68
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Who Experienced Single or Multiple Medical Encounters
Description: The number of subjects who experienced single or multiple encounters of medical events resulting in Emergency Department (ED) or hospitalization visits were reported
Time Frame: Within 6 months after any dose of MenACWY-CRM vaccination
Population: Analysis was performed on children, who received at least one dose of the study vaccine at a Kaiser Permanente Southern California (KPSC) facility.
Measure: Count of Participants; unit: Participants
Arm/Group | Exposure Group
Number analyzed (Participants) | 138
Participants
  Single medical encounter | 16
  Multiple medical encounters | 24

2. Primary Outcome: Number of Medical Encounters Following Any Dose of MenACWY-CRM Vaccination
Description: All medical encounters that required ED visits and hospitalizations within 6 months of vaccination were assessed. Medical encounters were considered pre-existing if all diagnoses made during an ED and/or hospitalization were pre-existing. If a study subject was first seen in the ED and subsequently transferred to the hospital, this was treated as a single episode of care.
Time Frame: Within 6 months after any dose of MenACWY-CRM
Population: as for outcome 1
Measure: Number; unit: Medical encounters
Arm/Group | Exposure Group
Number analyzed (Participants) | 138
Medical encounters
  ED and/or hospitalization encounters | 102
  Hospitalization only | 32
  Emergency department only | 57
  Emergency department to hospital transfer | 13

3. Primary Outcome: Incidence Rate of Medical Encounters Following Any Dose of MenACWY-CRM Vaccination
Description: The incidence rate of medical encounters was defined as the number of all captured encounters divided by the total person-time following MenACWY-CRM doses administered during the study period. The rate and Poisson 95% CI of medical encounters were calculated and presented as number per person-year. Person-time for each dose began at the date of the vaccination and ended at 6 months following vaccination, disenrollment, death, the end of data collection, or receipt of an additional dose of MenACWY-CRM, whichever came first.
Time Frame: Within 6 months after any dose of MenACWY-CRM
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Events per person-year
Arm/Group | Exposure Group
Number analyzed (Participants) | 138
Events per person-year
  Hospitalization only | 0.4 [0.3 to 0.5]
  Emergency department only | 0.6 [0.5 to 0.8]
  Emergency department to hospital transfer | 0.1 [0.1 to 0.3]

4. Primary Outcome: Number of Subjects Who Experienced Single or Mutiple Medical Diagnoses
Description: Number of subjects who experienced single or multiple medical diagnoses after the MenACWY-CRM dose were reported
Time Frame: Within 6 months after any dose of MenACWY-CRM
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Exposure Group
Number analyzed (Participants) | 138
Participants
  Single medical diagnosis | 6
  Multiple medical diganoses | 34

5. Primary Outcome: Number of Medical Diagnoses Following Any Dose of MenACWY-CRM Vaccination
Description: All medical diagnoses that required ED or hospitalization visits within 6 months of vaccination were assessed. Events with a history of the same diagnosis prior to the first dose of MenACWY-CRM vaccination were excluded as pre-existing conditions. Data presented for this outcome measure includes all medical diagnoses after the first and recurrent diagnoses. Diagnoses were identified from Electronic Medical Records (EMRs) of emergency and hospital care encounters by automated algorithm identification and then were manually reviewed by a physician to determine the final diagnosis/ diagnoses and diagnosis dates for the encounter. Diagnoses were classified according to International Classification of Diseases, ninth revision (ICD-9) codification. All medical diagnoses assessed are presented in short forms with the ICD code, due to character limitations.
Time Frame: Within 6 months after any dose of MenACWY-CRM
Population: as for outcome 1
Measure: Number; unit: Medical diagnoses
Arm/Group | Exposure Group
Number analyzed (Participants) | 138
Medical diagnoses
  Intestinal infection, other organism (ICD-008.8) | 2
  Septicemia, pseudomonas (038.43) | 1
  Pseudomonas infection (041.7) | 1
  Other specified bacterial infections(041.85) | 1
  Viral exanthem, unspecified(057.9) | 1
  Adenovirus infection(079.0) | 2
  Rhinovirus infection(079.3) | 1
  Other specified viral infection(079.89) | 2
  Unspecified viral infection(079.99) | 1
  Candidiasis of mouth(112.0) | 1
  Hyposmolality and/or hyponatremia(276.1) | 1
  Acidosis(276.2) | 2
  Dehydration(276.51) | 6
  Hyperpotassemia(276.7) | 1
  Hb-SS disease with crisis(282.62) | 2
  Other pancytopenia(284.19) | 1
  Acute posthemorrhagic anemia(285.1) | 1
  Anemia, unspecified(285.9) | 4
  Leukocytosis, unspecified(288.60) | 1
  Other specified delays in development(315.8) | 1
  Cerebral degeneration(331.7) | 1
  Epilepsy, unspecified(345.90) | 2
  Encephalopathy, unspecified(348.30) | 1
  Cerebral edema(348.5) | 1
  Conjunctivitis, unspecified(372.30) | 2
  Redness or discharge of eye(379.93) | 1
  Unspecified otitis media(382.9) | 6
  Cardiomegaly(429.3) | 1
  Subdural hemorrhage(432.1) | 1
  Cerebral artery occlusion(434.91) | 1
  Acute venous embolism and thrombosis(453.41) | 1
  Acute sinusitis, unspecified(461.9) | 1
  Acute upper respiratory infections(465.9) | 10
  Acute bronchitis(466.0) | 3
  Acute bronchiolitis,RSV(466.11) | 1
  Acute bronchiolitis,other organisms(466.19) | 1
  Chronic rhinitis(472.0) | 1
  Pneumonia, parainfluenza virus(480.2) | 2
  Pneumonia,other virus not classified(480.8) | 2
  Pneumococcal pneumonia(481) | 1
  Pneumonia, Pseudomonas(482.1) | 1
  Pneumonia, other gram-negative bacteria(482.83) | 1
  Pneumonia, mycoplasma pneumoniae(483.0) | 1
  Pneumonia, organism unspecified(486) | 5
  Influenza-other respiratory manifestations(487.1) | 4
  Asthma, unspecified type, unspecified(493.90) | 1
  Effusion, other (except tuberculous)(511.89) | 1
  Pulmonary congestion and hypostasis(514) | 1
  Unspecified pneumonopathy(516.9 | 1
  Pulmonary collapse(518.0) | 1
  Acute respiratory failure(518.81) | 3
  Other pulmonary insufficiency(518.82) | 2
  Other gastrostomy complications(536.49) | 1
  Other disorders-stomach & duodenum(537.89) | 1
  Noninfectious gastroenteritis &colitis,other(558.9 | 3
  Constipation, unspecified(564.00) | 2
  Anal sphincter tear (healed) (old)(569.43) | 1
  Urinary tract infection, site not specified(599.0) | 2
  Microscopic hematuria(599.72) | 1
  Diaper or napkin rash(691.0) | 3
  Allergic urticaria(708.0) | 1
  Pain in joint, lower leg(719.46) | 1
  Pain in limb(729.5) | 1
  Swelling of limb(729.81) | 1
  Other anomalies of great veins(747.49) | 1
  Other anomalies of female genitalia(752.49) | 1
  Anomalies of skull and face bones(756.0) | 1
  Hypoxicischemic encephalopathy,unspecified(768.70) | 1
  Complex febrile convulsions(780.32) | 1
  Other convulsions(780.39) | 2
  Fever, unspecified(780.60) | 25
  Fever with conditions classified elsewhere(780.61) | 11
  Postvaccination fever(780.63) | 1
  Altered mental status(780.97) | 1
  Rash & other nonspecific skin eruption(782.1) | 2
  Feeding difficulties & mismanagement(783.3) | 1
  Tachycardia, unspecified(785.0) | 2
  Tachypnea(786.06) | 1
  Wheezing(786.07) | 2
  Other respiratory abnormalities(786.09) | 3
  Cough(786.2) | 5
  Abnormal chest sounds(786.7) | 1
  Nausea with vomiting(787.01) | 2
  Vomiting alone(787.03) | 1
  Flatulence,eructation & gas pain(787.3) | 1
  Diarrhea(787.91) | 4
  Other symptoms involving digestive system(787.99) | 1
  Splenomegaly(789.2) | 2
  Bacteremia(790.7) | 1
  Viremia, unspecified(790.8) | 5
  Other abnormal finding of lung field(793.19) | 2
  Abnormal results,pulmonary function(794.2) | 1
  Hypoxemia(799.02) | 2
  Subarachnoid hemorrhage following injury(852.00) | 1
  Subdural hemorrhage following injury(852.2) | 1
  Subdural hemorrhage unspecified(852.20) | 1
  Open wound of finger(s)(883.0) | 1
  Insect bite,nonvenomous of lower limb(916.4) | 1
  Contusion of chest wall(922.1) | 1
  Foreign body in digestive system,unspecified(938) | 1
  Head injury, unspecified(959.01) | 1
  Knee, leg, ankle, and foot injury(959.7) | 1
  Child abuse, unspecified(995.50) | 1
  Child physical abuse(995.54) | 2
  Vascular device,implant,graft,complications(996.74 | 1
  Body systems,complications,hypertension(997.91) | 1
  Other external cause status(E000.8) | 2
  Other activity(E029.9) | 2
  Traffic accident-passenger injury(E812.1) | 1
  Home accidents(E849.0) | 2
  Accidents occurring in unspecified place(E849.9) | 3
  Surgical operations & procedures, (E878.8) | 1
  Other procedures, complication(E879.8) | 1
  Accidental fall on/from other stairs/steps(E880.9) | 1
  Unspecified fall(E888.9) | 1
  Bite of nonvenomous arthropod(E906.4) | 1
  Accidents caused by cutting and piercing(E920.8) | 1
  Other accidents(E928.8) | 1
  Unspecified accident(E928.9) | 1

6. Primary Outcome: Incidence Rate of Medical Diagnoses Following Any Dose of MenACWY- CRM Vaccination
Description: The incidence rate of diagnoses was defined as the number of all captured diagnoses divided by the total person-time following MenACWY-CRM doses administered during the study period. The rate and Poisson 95% CI of medical diagnoses were calculated and presented as number per person-year.Person-time for each dose began at the date of the vaccination and ended at 6 months following vaccination, disenrollment, death, the end of data collection, or receipt of an additional dose of MenACWY-CRM, whichever came first. Diagnoses were classified according ICD-9 codification. All medical diagnoses assessed are presented in short forms with the ICD code, due to character limitations.
Time Frame: Within 6 months after any dose of MenACWY-CRM
Population: Analysis was performed on medical events collected from children, who received at least one dose of the study vaccine at a Kaiser Permanente Southern California (KPSC) facility.
Measure: Number (95% Confidence Interval); unit: Events per person-year
Arm/Group | Exposure Group
Number analyzed (Participants) | 138
Events per person-year
  Intestinal infection, other organism (ICD-008.8) | 0.0 [0.0 to 0.1]
  Septicemia, pseudomonas (038.43) | 0.0 [0.0 to 0.1]
  Pseudomonas infection(041.7) | 0.0 [0.0 to 0.1]
  Other specified bacterial infections(041.85) | 0.0 [0.0 to 0.1]
  Viral exanthem, unspecified(057.9) | 0.0 [0.0 to 0.1]
  Adenovirus infection(079.0) | 0.0 [0.0 to 0.1]
  Rhinovirus infection(079.3) | 0.0 [0.0 to 0.1]
  Other specified viral infection(079.89) | 0.0 [0.0 to 0.1]
  Unspecified viral infection(079.99) | 0.0 [0.0 to 0.1]
  Candidiasis of mouth(112.0) | 0.0 [0.0 to 0.1]
  Hyposmolality and/or hyponatremia(276.1) | 0.0 [0.0 to 0.1]
  Acidosis(276.2) | 0.0 [0.0 to 0.1]
  Dehydration(276.51) | 0.1 [0.0 to 0.2]
  Hyperpotassemia(276.7) | 0.0 [0.0 to 0.1]
  Hb-SS disease with crisis(282.62) | 0.0 [0.0 to 0.1]
  Other pancytopenia(284.19) | 0.0 [0.0 to 0.1]
  Acute posthemorrhagic anemia(285.1) | 0.0 [0.0 to 0.1]
  Anemia, unspecified(285.9) | 0.0 [0.0 to 0.1]
  Leukocytosis, unspecified(288.60) | 0.0 [0.0 to 0.1]
  Other specified delays in development(315.8) | 0.0 [0.0 to 0.1]
  Cerebral degeneration(331.7) | 0.0 [0.0 to 0.1]
  Epilepsy, unspecified(345.90) | 0.0 [0.0 to 0.1]
  Encephalopathy, unspecified(348.30) | 0.0 [0.0 to 0.1]
  Cerebral edema(348.5) | 0.0 [0.0 to 0.1]
  Conjunctivitis, unspecified(372.30) | 0.0 [0.0 to 0.1]
  Redness or discharge of eye(379.93) | 0.0 [0.0 to 0.1]
  Unspecified otitis media(382.9) | 0.1 [0.0 to 0.2]
  Cardiomegaly(429.3) | 0.0 [0.0 to 0.1]
  Subdural hemorrhage(432.1) | 0.0 [0.0 to 0.1]
  Cerebral artery occlusion(434.91) | 0.0 [0.0 to 0.1]
  Acute venous embolism & thrombosis(453.41) | 0.0 [0.0 to 0.1]
  Acute sinusitis, unspecified(461.9) | 0.0 [0.0 to 0.1]
  Acute upper respiratory infections(465.9) | 0.1 [0.1 to 0.2]
  Acute bronchitis(466.0) | 0.0 [0.0 to 0.1]
  Acute bronchiolitis, RSV(466.11) | 0.0 [0.0 to 0.1]
  Acute bronchiolitis, other organisms(466.19) | 0.0 [0.0 to 0.1]
  Chronic rhinitis(472.0) | 0.0 [0.0 to 0.1]
  Pneumonia-parainfluenza virus(480.2) | 0.0 [0.0 to 0.1]
  Pneumonia, other virus(480.8) | 0.0 [0.0 to 0.1]
  Pneumococcal pneumonia(481) | 0.0 [0.0 to 0.1]
  Pneumonia, Pseudomonas(482.1) | 0.0 [0.0 to 0.1]
  Pneumonia, gram-negative bacteria(482.83) | 0.0 [0.0 to 0.1]
  Pneumonia, mycoplasma pneumoniae(483.0) | 0.0 [0.0 to 0.1]
  Pneumonia, organism unspecified(486) | 0.1 [0.0 to 0.1]
  Influenza-other respiratory manifestations(487.1) | 0.0 [0.0 to 0.1]
  Asthma,unspecified type,unspecified(493.90) | 0.0 [0.0 to 0.1]
  Effusion,other except tuberculous(511.89) | 0.0 [0.0 to 0.1]
  Pulmonary congestion & hypostasis(514) | 0.0 [0.0 to 0.1]
  Parieto/alveolar pneumonopathy,other(516.9) | 0.0 [0.0 to 0.1]
  Pulmonary collapse(518.0) | 0.0 [0.0 to 0.1]
  Acute respiratory failure(518.81) | 0.0 [0.0 to 0.1]
  Other pulmonary insufficiency(518.82) | 0.0 [0.0 to 0.1]
  Other gastrostomy complications(536.49) | 0.0 [0.0 to 0.1]
  Other disorders-stomach & duodenum(537.89) | 0.0 [0.0 to 0.1]
  Noninfectious gastroenteritis&colitis,other(558.9) | 0.0 [0.0 to 0.1]
  Constipation, unspecified(564.00) | 0.0 [0.0 to 0.1]
  Anal sphincter tear (healed)(old)(569.43) | 0.0 [0.0 to 0.1]
  Urinary tract infection,site not specified(599.0) | 0.0 [0.0 to 0.1]
  Microscopic hematuria(599.72) | 0.0 [0.0 to 0.1]
  Diaper or napkin rash(691.0) | 0.0 [0.0 to 0.1]
  Allergic urticaria(708.0) | 0.0 [0.0 to 0.1]
  Pain in joint, lower leg(719.46) | 0.0 [0.0 to 0.1]
  Pain in limb(729.5) | 0.0 [0.0 to 0.1]
  Swelling of limb(729.81) | 0.0 [0.0 to 0.1]
  Other anomalies of great veins(747.49) | 0.0 [0.0 to 0.1]
  Other anomalies of female genitalia(752.49) | 0.0 [0.0 to 0.1]
  Anomalies of skull & face bones(756.0) | 0.0 [0.0 to 0.1]
  Hypoxicischemic encephalopathy,unspecified(768.70) | 0.0 [0.0 to 0.1]
  Complex febrile convulsions(780.32) | 0.0 [0.0 to 0.1]
  Other convulsions(780.39) | 0.0 [0.0 to 0.1]
  Fever, unspecified(780.60) | 0.3 [0.2 to 0.4]
  Fever with conditions classified elsewhere(780.61) | 0.1 [0.1 to 0.2]
  Postvaccination fever(780.63) | 0.0 [0.0 to 0.1]
  Altered mental status(780.97) | 0.0 [0.0 to 0.1]
  Rash & other nonspecific skin eruption(782.1) | 0.0 [0.0 to 0.1]
  Feeding difficulties & mismanagement(783.3) | 0.0 [0.0 to 0.1]
  Tachycardia,unspecified(785.0) | 0.0 [0.0 to 0.1]
  Tachypnea(786.06) | 0.0 [0.0 to 0.1]
  Wheezing(786.07) | 0.0 [0.0 to 0.1]
  Other respiratory abnormalities(786.09) | 0.0 [0.0 to 0.1]
  Cough(786.2) | 0.1 [0.0 to 0.1]
  Abnormal chest sounds(786.7) | 0.0 [0.0 to 0.1]
  Nausea with vomiting(787.01) | 0.0 [0.0 to 0.1]
  Vomiting alone(787.03) | 0.0 [0.0 to 0.1]
  Flatulence, eructation & gas pain(787.3) | 0.0 [0.0 to 0.1]
  Diarrhea(787.91) | 0.0 [0.0 to 0.1]
  Other symptoms-digestive system(787.99) | 0.0 [0.0 to 0.1]
  Splenomegaly(789.2) | 0.0 [0.0 to 0.1]
  Bacteremia(790.7) | 0.0 [0.0 to 0.1]
  Viremia,unspecified(790.8) | 0.1 [0.0 to 0.1]
  Other abnormal finding of lung field(793.19) | 0.0 [0.0 to 0.1]
  Abnormal results,pulmonary function study(794.2) | 0.0 [0.0 to 0.1]
  Hypoxemia(799.02) | 0.0 [0.0 to 0.1]
  Subarachnoid hemorrhage,consciousness(852.00) | 0.0 [0.0 to 0.1]
  Subdural hemorrhage following injury(852.2) | 0.0 [0.0 to 0.1]
  Subdural hemorrhage,consciousness(852.20) | 0.0 [0.0 to 0.1]
  Open wound of finger(s)(883.0) | 0.0 [0.0 to 0.1]
  Insect bite,nonvenomous of lower limb(916.4) | 0.0 [0.0 to 0.1]
  Contusion of chest wall(922.1) | 0.0 [0.0 to 0.1]
  Foreign body in digestive system,unspecified(938) | 0.0 [0.0 to 0.1]
  Head injury, unspecified(959.01) | 0.0 [0.0 to 0.1]
  Knee,leg,ankle & foot injury(959.7) | 0.0 [0.0 to 0.1]
  Child abuse, unspecified(995.50) | 0.0 [0.0 to 0.1]
  Child physical abuse(995.54) | 0.0 [0.0 to 0.1]
  Vascular device implant&graft,complications(996.74 | 0.0 [0.0 to 0.1]
  Body systems,hypertension,complications(997.91) | 0.0 [0.0 to 0.1]
  Other external cause status(E000.8) | 0.0 [0.0 to 0.1]
  Other activity(E029.9) | 0.0 [0.0 to 0.1]
  Traffic accident-passenger injury(E812.1) | 0.0 [0.0 to 0.1]
  Home accidents(E849.0) | 0.0 [0.0 to 0.1]
  Accidents occurring in unspecified place(E849.9) | 0.0 [0.0 to 0.1]
  Surgical operations & procedures(E878.8) | 0.0 [0.0 to 0.1]
  Specified procedures, complications(E879.8) | 0.0 [0.0 to 0.1]
  Accidental fall on/from other stairs/steps(E880.9) | 0.0 [0.0 to 0.1]
  Unspecified fall(E888.9) | 0.0 [0.0 to 0.1]
  Bite of nonvenomous arthropod(E906.4) | 0.0 [0.0 to 0.1]
  Accidents caused by cutting & piercing(E920.8) | 0.0 [0.0 to 0.1]
  Other accidents(E928.8) | 0.0 [0.0 to 0.1]
  Unspecified accident(E928.9) | 0.0 [0.0 to 0.1]

ADVERSE EVENTS:
Time Frame: Not applicable as adverse events were not monitored in this study.
Description: Adverse events were not monitored in this study as this is an Non-interventional study based on the secondary use of Kaiser Permanente Southern California (KPSC) electronic records. There was no assessment of AEs related to study vaccination as MenACWY-CRM vaccine was given as part of the clinical care at KPSC. Reporting of number and rate of medical diagnosis is from pre-existing records in these centers.
Arm/Group | Exposure Group
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2016-08-11): https://cdn.clinicaltrials.gov/large-docs/88/NCT02287688/Prot_000.pdf
  • Statistical Analysis Plan (2015-10-30): https://cdn.clinicaltrials.gov/large-docs/88/NCT02287688/SAP_001.pdf